CLINICAL TRIAL: NCT06629194
Title: Validation of Scoring Systems for Differentiating Intestinal Tuberculosis from Crohn's Disease Utilizing Clinical, Endoscopic, and Interferon-gamma Releasing Assay in Asian Population
Brief Title: Validation of Scoring Systems for Differentiating Intestinal Tuberculosis from Crohn's Disease
Status: Recruiting | Type: Observational
Sponsor: Mahidol University (Other)
Collaborators: Korean Association for the Study of Intestinal Diseases (Other)
Responsible Party: Principal Investigator, Julajak Limsrivilai, Assoc. Prof., Mahidol University
Other Study IDs: Si212/2024
Record Dates: First submitted 2024-06-09; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Crohn Disease; Intestinal Tuberculosis; Differential Diagnosis
Keywords: Intestinal tuberculosis; Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Crohn's disease: Patients who were diagnosed Crohn's disease
  - Diagnosis of Crohn's disease is based on clinical, endoscopic, pathological, and/or radiological findings which is confirmed by clinical & endoscopic response to Crohn's disease treatment
  Interventions: Diagnostic Test: interferon gamma releasing assay (IGRA)
- Intestinal tuberculosis: Patients who were diagnosed intestinal tuberculosis.
  * Criteria of intestinal tuberculosis diagnosis includes any of following:
    i. Presence of caseating granuloma on pathological examination of specimens ii. Presence of acid-fast bacilli on pathological examination of specimens iii. PCR positive for Mycobacterium tuberculosis iv. Tissue culture growing organisms consistent with Mycobacterium tuberculosis v. Negative results in i to iv but response to empirical treatment with antituberculous therapy
  * All are required to have clinical and endoscopic response to antituberculous therapy (ATT) treatment
  Interventions: Diagnostic Test: interferon gamma releasing assay (IGRA)

INTERVENTIONS:
Diagnostic Test: interferon gamma releasing assay (IGRA) — All patients who suspected CD or TB will be tested for interferon-gamma releasing assay. An interferon-gamma release assay is a blood test that measures the body's immune response to Mycobacterium tuberculosis, the bacteria that causes tuberculosis.

SUMMARY:
Differentiating CD from intestinal tuberculosis (ITB) is difficult due to the low sensitivities of currently available diagnostic tests. The Asia-Pacific guideline recommends anti-tuberculous therapy (ATT) for 8-12 weeks in patients with diagnostic uncertainty due to the risk of disseminated tuberculosis if patients with ITB are misdiagnosed with CD, and are prescribed immunosuppressive therapy. However, treatment with ATT has many side effects and may delay treatment in patients with CD, and this may cause severe relapse and developing complications. Many studies found that some clinical, endoscopy, pathology, radiology, and serology findings can help to improve diagnostic accuracy in these patients. However, no single diagnostic parameter can distinguish between CD and ITB. As a result, many models were developed that include various factors and modalities, and many of those models have been reported to have high performance. However, the number of studies performed to validate those models externally was limited. Correspondingly, this study is designed to prospectively validate models that integrate more advanced parameters (e.g., IGRA, CT enterography findings) with clinical, endoscopic, or pathological findings. However, it aims mainly to evaluate the model integrating clinical, endoscopic, and serological variables since CT enterography and pathological interpretation require experienced radiologists and pathologists but they are not available in many centers.

DETAILED DESCRIPTION:
Crohn's disease (CD) incidence has been increasing in Asia over the last few decades [1]. Moreover, differentiating CD from intestinal tuberculosis (ITB) is difficult due to the low sensitivities of currently available diagnostic tests. The 5.3- 37.5% sensitivity of acid-fast bacilli (AFB) specimen staining, the 23%-46% sensitivity of mycobacterial culture, and the 36.4-67.9% sensitivity of tissue polymerase chain reaction (PCR) are all too low to confidently distinguish between these two conditions and exclude a diagnosis of ITB. The Asia-Pacific guideline recommends anti-tuberculous therapy (ATT) for 8-12 weeks in patients with diagnostic uncertainty due to the risk of disseminated tuberculosis if patients with ITB are misdiagnosed with CD, and are prescribed immunosuppressive therapy. However, treatment with ATT has many side effects and may delay treatment in patients with CD, and this may cause severe relapse and developing complications. In response, many studies were conducted to identify and classify characteristics that can help to distinguish between these two diseases. Those studies found that some clinical, endoscopy, pathology, radiology, and serology findings can help to improve diagnostic accuracy in these patients. However, no single diagnostic parameter can distinguish between CD and ITB. As a result, many models were developed that include various factors and modalities, and many of those models have been reported to have high performance. However, the number of studies performed to externally validate those models was limited.

To address this inadequacy, J Limsrivilai, et al. conducted a multicenter retrospective study comparing the ability of each different diagnostic model consisting of different combinations of basic clinical, endoscopic, and pathologic parameters affordable to resource-limited healthcare settings at differentiating CD and ITB patients. In the study, several differentiating models were included and applied to a cohort of 590 patients from Thailand and Hong Kong to validate the models. The results from the study concluded that the accuracy of a differentiating model is directly correlated with the number of diagnostic modalities and variables of the model with the ITBvsCD-CEP model, which includes 22 variables from clinical, endoscopy, and pathology parameters, demonstrating the highest AUROC as high as 0.887. Although the model demonstrated such impressive diagnostic ability, its application in real-life clinical practice has remained controversial as around 10% of ITB patients would still be misdiagnosed and thus receive the wrong treatments. Integrating more diagnostic modalities, such as interferon gamma-releasing assay (IGRA) and CT enterography, may be helpful.

Correspondingly, this study is designed to prospectively validate models that integrate more advanced parameters (e.g., IGRA, CT enterography findings) with clinical, endoscopic, or pathological findings. However, it aims mainly to evaluate the model integrating clinical, endoscopic, and serological variables since CT enterography and pathological interpretation require experienced radiologists and pathologists but they are not available in many centers.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ages 18 years or older
2. Undergoing colonoscopy and found ileal or colonic ulcers
3. Have ileal and/or colonic tissue sent for mycobacterial tests, including stain for AFB, PCR, and culture
4. Diagnosed with either intestinal tuberculosis or Crohn's disease a. Criteria of intestinal tuberculosis diagnosis includes any of following: i. Presence of caseating granuloma on pathological examination of specimens ii. Presence of acid-fast bacilli on pathological examination of specimens iii. PCR positive for Mycobacterium tuberculosis iv. Tissue culture growing organisms consistent with Mycobacterium tuberculosis v. Negative results in i to iv but response to empirical treatment with antituberculous therapy All are required to have clinical and endoscopic response to antituberculous therapy (ATT) treatment b. Diagnosis of Crohn's disease is based on clinical, endoscopic, pathological, and/or radiological findings which is confirmed by clinical & endoscopic response to Crohn's disease treatment

Exclusion Criteria:

1. Patients with ileal/colonic ulcers caused by other diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who had clinical symptoms suspicious of either Crohn's disease or intestinal tuberculosis are eligible.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2024-06-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the ITBvsCD model | with 4 weeks of colonoscopy
  The ITBvsCD model performance in differentiating Crohns disease from intestinal tuberculosis will be evaluated by area under the receiver operating characteristic (ROC) curve.

CONTACTS AND LOCATIONS:
Overall Officials: Julajak Limsrivilai, Principal Investigator — Division of Gastroenterology, Department of Medicine, Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Thailand
Locations (2):
- Thailand (2):
  - Assoc. Prof. Julajak Limsrivilai, MD, Bangkok Noi, Bangkok
  - Gastroenterology division, Faculty of Medicine, Siriraj Hospital, Mahidol University, Bangkok

IPD SHARING:
Plan to Share IPD: No